CLINICAL TRIAL: NCT00185913
Title: Identification of Serum Markers For Tumor Hypoxia in Non-Small Cell Lung Cancers
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Quynh-Thu Le, Stanford University School of Medicine
Other Study IDs: LUN0006; 75318; LUN0006; NCT00185913
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2010-04-22 (Estimated); Status verified 2010-04

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood

SUMMARY:
The purpose of the study is to identify a surrogate serum marker for tumor hypoxia in patients with lung cancers.

ELIGIBILITY:
Inclusion Criteria:- Newly diagnosed patients with lung cancer who are undergoing surgical resection of their tumors Exclusion Criteria:- Patients without non-small cell lung cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed patients with lung cancer who are undergoing surgical resection of their tumors
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2000-09; Primary Completion 2003-10 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Quynh-Thu Le, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States